CLINICAL TRIAL: NCT03996135
Title: Study of the Effectiveness of a Venous Illumination System for Peripheral Venous Pathways in Cirrhotic Patients
Brief Title: Evaluation of Accuvein in Cirrhotics Patients
Acronym: CIRRVVUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-043
Record Dates: First submitted 2019-06-05; First posted 2019-06-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : Cannulation with AccuVein AV400 (Experimental): Cirrhotic patients benefit from the support of a venous illumination device for each peripheral venous cannulation
  Interventions: Device: Cannulation with AccuVein AV400
- Control (No Intervention): Cirrhotic patients benefit from the standard technique of peripheral veinous catheter placement.

INTERVENTIONS:
Device: Cannulation with AccuVein AV400 — Cannulation using AccuVein AV400 device
  Other Names: AccuVein AV400
  Arms: Experimental : Cannulation with AccuVein AV400

SUMMARY:
The objective of this study is to evaluate the effectiveness of AccuVein AV400 to facilitate placement of peripheral intravenous catheters in cirrhotic adults by comparing the success rate of the first attempt to install a peripheral venous catheter with or without AccuVein AV400®.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient presenting a liver cirrhosis
* Patient requiring the placement of a venous peripheral catheter
* Patient informed and giving free and informed consent
* Patient affiliated to a French social security scheme

Exclusion Criteria:

* Patient under 18 years old
* Patient unable to give consent
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
First Attempt Success Rate of Cannulation | baseline
  Firt attempt success of positional for each peripheral venous catheter and expressed as a percentage in cirrhotic patients during hospitalization.

SECONDARY OUTCOMES:
change of the score A-DIVA | baseline and end of hospitalization (up to a month)
  Scores A-DIVA between beginning and end of hospitalization between the two groups
Cost | baseline
  Cost of consumables used in euro between the two groups
Life expectancy of the catheter | baseline
  Life expectancy of the catheter between the two groups
Utilisation of a central venous catheter | baseline
  Use of a central venous catheter (y/n)
Pain's score | baseline
  visual analogic scale
Numbers of attempts | baseline
  Number of attempts between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France